CLINICAL TRIAL: NCT07122219
Title: Enhancing Uptake of Needle and Syringe Programs in Canadian Federal Prisons
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Collaborators: Yale University (Other); Burnet Institute (Other); Kirby Institute (Other Government)
Responsible Party: Principal Investigator, Nadine Kronfli, Nominated Principal Investigator, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: 2023-9201; 195710 (Other Grant/Funding Number: Canadian Institutes of Health Research)
Record Dates: First submitted 2025-08-07; First posted 2025-08-14 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: HIV; Hepatitis C Virus (HCV)
Keywords: Needle-Exchange Programs; Prisons; Health Services for Prisoners; Blood-Borne Pathogens; HIV; Hepatitis C
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Intervention Model Description: Hybrid type 2 stepped-wedge implementation trial. All sites will receive the intervention (NIATx); the order in which they receive the intervention was non-randomized*.
  *Originally randomized; allocation was modified due to logistical constraints
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- NIATx group 1 (Experimental): Control (month 1-6) then NIATx (month 7-30) then Maintenance (month 31-42)
  Interventions: Behavioral: NIATx
- NIATx group 2 (Experimental): Control (month 7-12) then NIATx (month 13-36) then Maintenance (month 37-48)
  Interventions: Behavioral: NIATx
- NIATx group 3 (Experimental): Control (month 13-18) then NIATx (month 19-42) then Maintenance (month 43-54)
  Interventions: Behavioral: NIATx

INTERVENTIONS:
Behavioral: NIATx — The Network for the Improvement of Addiction Treatment (NIATx) model uses a bundle of implementation tools that include expert facilitation (coaching) and quality process improvement specifically for behavioural healthcare settings to improve access and retention in treatment.

SUMMARY:
This study is focused on improving the implementation of Prison Needle Exchange Programs (PNEPs) in Canadian federal prisons, with the goal of increasing the uptake of these programs among people who inject drugs in prison. The study is being conducted in nine federal prisons, including five women's prisons, where a higher proportion of incarcerated individuals report a history of injection drug use. This study aims to improve PNEP adoption and sustainability by identifying barriers and facilitators and implementing evidence-based strategies to enhance program engagement.

DETAILED DESCRIPTION:
Using a step-wedge design, we will conduct a Type 2 hybrid implementation trial to assess the extent to which PNEP uptake is improved over 24 months of observation using the Network for the Improvement of Addiction Treatment (NIATx) implementation strategy bundle. Nine prisons were non-randomly* allocated to one of three groups, with the groups receiving the intervention (i.e., NIATx) over 24 months at staggered time intervals (every 6 months). This will be followed by an additional 12 month post-intervention period, when sustainability will be assessed.

*Originally randomized; allocation was modified due to logistical constraints

ELIGIBILITY:
Inclusion Criteria:

* All people incarcerated at a study site during the intervention period

Exclusion Criteria:

- None (site level intervention)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 548 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2028-02-29 (Estimated); Study Completion 2029-09-30 (Estimated)

PRIMARY OUTCOMES:
Effectiveness | From start to end of intervention period (24 months)
  Number of participants on the PNEP

SECONDARY OUTCOMES:
Bloodborne virus cascade of care | From start to end of intervention period (24 months)
  Number of HIV and hepatitis C virus screenings/tests, diagnoses, and treatment initiations, among the total prison population
Enrollment in opioid agonist therapy | From start to end of intervention period (24 months)
  The number of people who inject drugs who access opioid agonist therapy among the total prison population

CONTACTS AND LOCATIONS:
Overall Officials: Nadine Kronfli, Principal Investigator — Research Institute of the McGill University Health Centre; Frederick L. Altice, Principal Investigator — Yale University
Locations (9):
- Canada (9):
  - Edmonton Institution for Women, Edmonton, Alberta
  - Fraser Valley Institution for Women, Abbotsford, British Columbia
  - Mission Institution, Mission, British Columbia
  - Dorchester Medium, Dorchester, New Brunswick
  - Atlantic Institution, Smiths Crossing, New Brunswick
  - Nova Institution for Women, Truro, Nova Scotia
  - Joyceville Institution, Kingston, Ontario
  - Grand Valley Institution for Women, Kitchener, Ontario
  - Joliette Institution for Women, Joliette, Quebec

IPD SHARING:
Plan to Share IPD: No
Data requests can be made to Correctional Service Canada